CLINICAL TRIAL: NCT02530385
Title: Placebo Controlled Study of Fecal Microbiota Transplant (FMT) to Impact Body Weight and Glycemic Control in Adults Using a Frozen Encapsulated Inoculum
Brief Title: Fecal Microbiota Transplant for Improvement of Metabolism
Acronym: FMT-TRIM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elaine W. Yu, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-P001632
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- FMT (Experimental): Active FMT capsules
  Interventions: Biological: FMT Capsules
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Other: Placebo Capsules

INTERVENTIONS:
Other: Placebo Capsules — Placebo capsules contain powdered cocoa and gelatin
  Arms: Placebo
Biological: FMT Capsules — Capsules will be generated as per FDA-approved procedures
  Arms: FMT

SUMMARY:
The purpose of this study is to study the impact of gut bacteria on weight. Fecal microbiota transplantation (FMT) transfers intestinal bacteria by a "stool transplant" from a healthy, lean person to a person with obesity.

DETAILED DESCRIPTION:
Multiple lines of evidence suggest that gut microbiota play an important role in regulating human metabolism. In this study, subjects will receive FMT capsules from lean metabolically healthy donors to study effects on body weight and insulin sensitivity. Subjects who participate will be randomized 1:1 to receive either active FMT capsules or placebo capsules. Subjects and providers will be blinded to treatment assignment. The study will last for 24 weeks. Subjects will be asked to come to MGH for a baseline visit at week 0, return for 6 weekly visits and come back at week 12. Major study outcomes include change in weight, insulin sensitivity, and body composition. Fecal samples will also be collected for intestinal microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 kg/m2
* Because of frequent study mandated visits, only subjects living within reasonable driving distance of Massachusetts General Hospital may be enrolled

Exclusion Criteria:

* Pregnant women
* Use of diabetic medications or weight loss medications in the preceding 1 year
* Significant gastrointestinal disorders
* Significant food allergies
* Immunosuppressed patients

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Yu EW, Gao L, Stastka P, Cheney MC, Mahabamunuge J, Torres Soto M, Ford CB, Bryant JA, Henn MR, Hohmann EL. Fecal microbiota transplantation for the improvement of metabolism in obesity: The FMT-TRIM double-blind placebo-controlled pilot trial. PLoS Med. 2020 Mar 9;17(3):e1003051. doi: 10.1371/journal.pmed.1003051. eCollection 2020 Mar. PMID 32150549

RESULTS

PARTICIPANT FLOW:
Groups:
- FMT Capsules: Active FMT capsules
  FMT Capsules: Capsules will be generated as per FDA-approved procedures
Period: Overall Study
Arm/Group | Placebo | FMT Capsules
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMT Capsules | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (8.4) | 38.5 (8.8) | 40.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Insulin Resistance Based on Insulin-Stimulated Glucose Uptake (M) During Hyperinsulinemic Euglycemic Clamp
Time Frame: Baseline and 6 weeks
Population: 2 participants in the FMT Capsules group did not complete the 6 week study visit: 1 withdrew prior to the visit; 1 missed due to a scheduling issue.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | FMT Capsules
Number analyzed (Participants) | 12 | 10
percent change | -3 (32) | 5 (12)
Statistical Analysis 1: Comparison: Placebo vs FMT Capsules; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Insulin Resistance Based on Homeostasic Model Assessment of Insulin Resistance (HOMA-IR)
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Placebo | FMT Capsules
Number analyzed (Participants) | 12 | 12
unitless
  Baseline | 3.5 (1.9) | 3.5 (1.4)
  12 weeks | 4.8 (1.7) | 4.7 (2.0)
Statistical Analysis 1: Comparison: Placebo vs FMT Capsules; Test type: Superiority; p = 0.70, Mixed Models Analysis

3. Secondary Outcome: Body Weight (Metabolic Scale)
Description: Change in body weight from baseline to 12 weeks will be measured on a metabolic scale.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | FMT Capsules
Number analyzed (Participants) | 12 | 12
kg
  Baseline | 111 (20) | 110 (26)
  12 weeks | 111 (19) | 111 (27)
Statistical Analysis 1: Comparison: Placebo vs FMT Capsules; Test type: Superiority; p = 0.93, Mixed Models Analysis

4. Secondary Outcome: Lean Mass
Description: Change in lean mass from baseline to 12 weeks measured via dual-energy x-ray absorptiometry
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | FMT Capsules
Number analyzed (Participants) | 12 | 12
kg
  Baseline | 58 (12) | 60 (15)
  12 week | 58 (11) | 61 (16)
Statistical Analysis 1: Comparison: Placebo vs FMT Capsules; Test type: Superiority; p = 0.90, Mixed Models Analysis

5. Secondary Outcome: Fat Mass
Description: Change in fat mass from baseline to 12 weeks measured via dual-energy x-ray absorptiometry
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | FMT Capsules
Number analyzed (Participants) | 12 | 12
kg
  Baseline | 53 (10) | 49 (13)
  12 weeks | 52 (10) | 50 (14)
Statistical Analysis 1: Comparison: Placebo vs FMT Capsules; Test type: Superiority; p = 0.32, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Questionnaire administered at every study visit.
Arm/Group | Placebo | FMT Capsules
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | FMT Capsules (N=12)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | FMT Capsules (N=12)
Fever (General disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 10
Bloating/Abdominal Pain (Gastrointestinal disorders) | 5 | 7
Nausea/Vomiting (Gastrointestinal disorders) | 6 | 6
Fatigue (General disorders) | 3 | 5
Headache (General disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT02530385/Prot_SAP_000.pdf